CLINICAL TRIAL: NCT02135042
Title: Randomized Phase II and Phase III Studies of Individualized Treatment for Nasopharyngeal Carcinoma Based on Biomarker Epstein Barr Virus (EBV) Deoxyribonucleic Acid (DNA)
Brief Title: Individualized Treatment in Treating Patients With Stage II-IVB Nasopharyngeal Cancer Based on EBV DNA
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-HN001; NCI-2014-00635 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN001 (Other: NRG Oncology); NRG-HN001 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH); NCT02179164 (obsolete NCT alias)
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Epstein-Barr Virus Infection; Stage II Nasopharyngeal Carcinoma; Stage III Nasopharyngeal Carcinoma; Stage IVA Nasopharyngeal Carcinoma; Stage IVB Nasopharyngeal Carcinoma
MeSH Terms: conditions — Epstein-Barr Virus Infections; Nasopharyngeal Carcinoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Watchful Waiting; Fluorouracil; dehydroftorafur; Gemcitabine; Radiotherapy, Intensity-Modulated; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (chemoradiation, cisplatin, fluorouracil) (Active Comparator): Patients receive PF regimen comprising cisplatin IV over 60-120 minutes and fluorouracil IV over 96 hours continuously beginning at least 4 weeks after completion of IMRT. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Arm II (chemoradiation, gemcitabine hydrochloride, paclitaxel) (Experimental): Patients receive GT regimen comprising paclitaxel IV over 1 hour and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 at least 4 weeks after completion of IMRT. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Arm III (chemoradiation, cisplatin, fluorouracil) (Active Comparator): Patients receive PF regimen as in Arm I of Phase II.
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Arm IV (chemoradiation, observation) (Experimental): Patients undergo clinical observation.
  Interventions: Drug: Cisplatin; Other: Clinical Observation; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Other: Clinical Observation — Undergo clinical observation
  Arms: Arm IV (chemoradiation, observation)
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Actino-Hermal; Adrucil; Arumel; Cytosafe; Efudex; Efurix; Fiverocil; Fluoro Uracil; Fluoroplex; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Flurox; Ribofluor; Ro 2-9757; Ro-2-9757; Timazin
  Arms: Arm I (chemoradiation, cisplatin, fluorouracil); Arm III (chemoradiation, cisplatin, fluorouracil)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
  Arms: Arm II (chemoradiation, gemcitabine hydrochloride, paclitaxel)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm II (chemoradiation, gemcitabine hydrochloride, paclitaxel)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
There are two study questions we are asking in this randomized phase II/III trial based on a blood biomarker, Epstein Barr virus (EBV) deoxyribonucleic acid (DNA) for locoregionally advanced non-metastatic nasopharyngeal cancer. All patients will first undergo standard concurrent chemotherapy and radiation therapy. When this standard treatment is completed, if there is no detectable EBV DNA in their plasma, then patients are randomized to either standard adjuvant cisplatin and fluorouracil chemotherapy or observation. If there is still detectable levels of plasma EBV DNA, patients will be randomized to standard cisplatin and fluorouracil chemotherapy versus gemcitabine and paclitaxel. Radiation therapy uses high energy x rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, fluorouracil, gemcitabine hydrochloride, and paclitaxel work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving cisplatin and fluorouracil is more effective than gemcitabine hydrochloride and paclitaxel after radiation therapy in treating patients with nasopharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether substituting adjuvant concurrent high dose cisplatin (CDDP) and fluorouracil (5-FU) with gemcitabine (gemcitabine hydrochloride) and paclitaxel will result in superior progression-free survival. (Detectable Plasma Epstein Barr Virus [EBV] Deoxyribonucleic Acid [DNA] Cohort randomized Phase II) II. To determine whether omitting adjuvant CDDP and 5-FU (observation alone in the adjuvant setting) will result in non-inferior overall survival as compared with those patients receiving adjuvant CDDP and 5-FU chemotherapy. (Undetectable Plasma EBV DNA Cohort Phase III)

SECONDARY OBJECTIVES:

I. Time to distant metastasis. (Randomized Phase II and Phase III) II. Time to local progression. (Randomized Phase II and Phase III) III. Time to regional progression. (Randomized Phase II and Phase III) IV. Progression-free survival (Undetectable Cohort). V. Overall survival (Detectable Cohort). VI. Acute and late toxicity profiles based on clinician-reported Common Terminology Criteria for Adverse Events (CTCAE), version (v.) 4. (Randomized Phase II and Phase III) VII. Death during or within 30 days of end of protocol treatment. (Randomized Phase II and Phase III) VIII. Quality of life (general and physical well-being). (Randomized Phase II and Phase III) IX. Quality of life (hearing). (Randomized Phase II and Phase III) X. Quality of life (peripheral neuropathy). (Randomized Phase II and Phase III) XI. Cost effectiveness. (Randomized Phase II and Phase III)

OUTLINE:

Patients undergo intensity modulated radiation therapy (IMRT) once daily (QD) 5 days a week for 6.5 weeks and receive low-dose cisplatin intravenously (IV) over 30-60 minutes once weekly during IMRT. Beginning 1 week after chemoradiation, plasma samples are collected for EBV DNA analysis.

PHASE II: Patients with detectable EBV DNA from pre-treatment analysis are randomized to 1 of 2 treatment arms.

ARM I: Patients receive PF regimen comprising cisplatin IV over 60-120 minutes and fluorouracil IV over 96 hours continuously beginning at least 4 weeks after completion of IMRT. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive GT regimen comprising paclitaxel IV over 1 hour and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 at least 4 weeks after completion of IMRT. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

PHASE III:

Patients with undetectable EBV DNA from pre-treatment analysis are randomized to 1 of 2 treatment arms.

ARM III: Patients receive PF regimen as in Arm I.

ARM IV: Patients undergo clinical observation.

After completion of study treatment, patients are followed up every 4 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven (from primary lesion and/or lymph nodes) diagnosis of cancer of the nasopharynx
* Sites are required to complete Step 1 registration before submitting specimens for EBV DNA analysis.

  * Patients must have detectable pretreatment plasma EBV DNA, determined by the central lab prior to Step 2 registration (see Section 10.2 for details of specimen submission).
  * For patients who have detectable plasma EBV DNA tested at one of the credentialed central labs (listed on the EBV DNA Testing Specimen Transmittal form) within 28 days prior to Step 1 registration: that test result can be used for eligibility without the need for re-testing. To use this test result for eligibility, the central lab must enter the test result through the pathology portal, and the site must follow the instructions in Section 5.4.
* Stage II-IVB disease (AJCC, 7th ed.) with no evidence of distant metastasis, based upon the following minimum diagnostic workup:

  * History/physical examination by a Medical Oncologist or Clinical Oncologist or Radiation Oncologist or ENT, which must include an endoscopic evaluation, a complete list of current medications, and assessment of weight and weight loss in the past 6 months within 21 days prior to registration;
  * Evaluation of tumor extent required within 28 days prior to registration:
* MRI of the nasopharynx and neck; or CT of the nasopharynx and neck with ≤ 3 mm contiguous slices with contrast and bone windows (to evaluate base of skull involvement).

Note: If a treatment planning CT scan is used, it must be with ≤ 3 mm contiguous slices with contrast and be read by a radiologist.

Please refer to section 6.3.2 for MRI requirement for target delineation.

* To rule out distant metastasis, patients must undergo the following imaging within 28 days prior to registration:

  1. a CT scan with contrast of the chest and abdomen (required), and the pelvis (optional), or a total body PET/CT scan (non-contrast PET/CT is acceptable);
  2. a bone scan only when there is suspicion of bone metastases (a PET/CT scan can substitute for the bone scan).
* Zubrod performance status 0-1 within 21 days prior to registration
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 8.0 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] ≥ 8.0 g/dl is acceptable)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 x institutional ULN
* Alkaline phosphatase ≤ 1.5 x institutional ULN
* Serum creatinine ≤ 1.5 mg/dl or calculated creatinine clearance (CC) ≥ 50 ml/min determined by 24-hour urine collection or estimated by Cockcroft-Gault formula
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential
* Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control throughout protocol treatment
* Patient must provide study specific informed consent prior to study entry, including the mandatory pre-treatment plasma EBV DNA assay

Exclusion Criteria:

* Prior invasive malignancy (except node negative, non-melanomatous skin cancer) unless disease free for a minimum of 1095 days (3 years) (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable; however, at least 6-weeks recovery is necessary if the last regimen included nitrosourea or mitomycin
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Patients with hearing loss assessed to be primarily sensorineural in nature, requiring a hearing aid, or intervention (i.e. interfering in a clinically significant way with activities of daily living); a conductive hearing loss that is tumor-related is allowed
* ≥ Grade 2 peripheral sensory neuropathy (CTCAE, v. 4.0)
* Severe, active co-morbidity, defined as follows:

  * Major medical or psychiatric illness, which in the investigator's opinion would interfere with the completion of therapy and follow up or with full understanding of the risks and potential complications of the therapy
  * Unstable angina and/or uncontrolled congestive heart failure within the past 6 months
  * Myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; note that patients switched from IV antibiotics and currently on oral antibiotics whose infection is assessed to be adequately treated or controlled are eligible
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that Human Immunodeficiency Virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Prior allergic reaction to the study drug(s) involved in this protocol
* Patients with undetectable pre-treatment plasma EBV DNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2014-04-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) (Undetectable Plasma EBV DNA Cohort Phase III) | Up to 7 years
  Estimated using the Kaplan-Meier method for each arm. Their distributions will be compared between treatment arms with a 1-sided log rank test. The confidence interval approach will be used for the final analysis of OS.
Progression-free survival (PFS) (Detectable Plasma EBV DNA Cohort Phase II) | Up to 7 years
  Estimated using the Kaplan-Meier method for each arm. Their distributions will be compared between treatment arms with a 1-sided log rank test. A one-sided log rank test will be used to compare the PFS at a significance level of 0.1379.

SECONDARY OUTCOMES:
Changes in pure tone audiometry (Phase II and III) | Baseline to up to 1 year
  Correlation between categorical measures will be summarized by odds ratios, chi-square tests, and associated measures. Adjusted correlation may be derived from analysis of covariance (ANCOVA) models or derived directly using nonparametric analysis of variance (ANOVA) models if normality assumption is violated. Correlations between HHIE-S PRO scores and PTA and FACT-NP hearing, and PTA will be compared as dependent statistics
Changes in QOL (hearing) as assessed by the Hearing Handicap Inventory for the Elderly-Screening version (HHIE-S) (Phase II and III) | Baseline to up to 24 months
  QOL analysis including overall score and change from baseline will be summarized using mean and standard deviation at each time point for each arm. Overall and nasopharyngeal-specific QOL, hearing QOL (FACT-NP hearing domain, HHIE-S scores), peripheral neuropathy QOL over the short and long term and pure-tone audiometry (PTA) scores will be compared using a two sample independent t test and paired t test if the comparison is within the experimental arm between different time points.
Changes in QOL (peripheral neuropathy) as assessed by the FACT-Taxane (Phase II and III) | Baseline to up to 24 months
Changes in quality of life (QOL) (general and physical well-being) assessed using the Functional Assessment of Cancer Therapy (FACT)-Nasopharyngeal (NP) (Phase II and III) | Baseline to up to 24 months
  Changes in patient reported outcome (PRO) scores will be correlated to clearance or non-clearance of EBV titers. Descriptive statistics derived from FACT-NP will be used to enrich the understanding of QOL as it pertains to the 2 phase III arms of observation versus additional adjuvant chemotherapy. Univariable and multivariable analysis will be performed using the Cox proportional hazards model for OS and distant metastasis. Pearson correlation will be estimated between general and physical well-being. QOL measures and change from baseline will be correlated to EBV DNA.
Cost effectiveness as assessed by the health-related QOL (HRQOL) from the EuroQol (EQ-5D) instrument (Phase II and III) | Up to 24 months
  Incremental cost effectiveness ratios will be compared to determine the probability of cost effectiveness of various interventions, with sensitivity analyses to identify model weaknesses. The expected value of perfect information will be determined to delimit the upper boundary for cost-effective future investment in this area of research.
Incidence of acute grade 3-5 adverse events (Phase II and III) | Up to 7 years
  Rates of specific acute toxicity profiles and late toxicity profiles will be estimated using a binomial distribution along with their associated 95% confidence intervals and will be compared using Fisher's exact test between the 2 treatment arms.
Incidence of death (Phase II and III) | Up to 30 days of end of protocol treatment
Incidence of late grade 3-5 adverse events (Phase II and III) | Up to 7 years
  Rates of specific acute toxicity profiles and late toxicity profiles will be estimated using a binomial distribution along with their associated 95% confidence intervals and will be compared using Fisher's exact test between the 2 treatment arms.
OS (Detectable Plasma EBV DNA Cohort Phase II) | Up to 7 years
  Estimated using the Kaplan-Meier method for each arm. Their distributions will be compared between treatment arms with a 1-sided log rank test.
PFS (Undetectable Plasma EBV DNA Cohort Phase III) | Up to 7 years
  Estimated using the Kaplan-Meier method for each arm. Their distributions will be compared between treatment arms with a 1-sided log rank test.
Time to distant metastasis (DM) (Phase II and III) | Up to 7 years
  The cumulative incidence method will be used to estimate local, regional, and distant failure rates. The failure rates for the experimental treatment will be compared against the control using a failure-specific log-rank test. Multivariate analysis will be performed using the Cox proportional hazards model.
Time to local progression (Phase II and III) | Up to 7 years
  The cumulative incidence method will be used to estimate local, regional, and distant failure rates. The failure rates for the experimental treatment will be compared against the control using a failure-specific log-rank test. Multivariate analysis will be performed using the Cox proportional hazards model.
Time to regional progression (Phase II and III) | Up to 7 years
  Defined as an estimated increase in the size of the tumor (product of the perpendicular diameters of the two largest dimensions) of greater than 25%, taking as reference the smallest value of all previous measurements or appearance of new areas of malignant disease. The cumulative incidence method will be used to estimate local, regional, and distant failure rates. The failure rates for the experimental treatment will be compared against the control using a failure-specific log-rank test. Multivariate analysis will be performed using the Cox proportional hazards model.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, Principal Investigator — NRG Oncology
Locations (215):
- United States (199):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Fresno Cancer Center, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - SCL Health Cancer Centers of Colorado - Lutheran Medical Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Yale University, New Haven, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - New York Proton Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Cleveland Clinic Akron General, Akron, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- China (3):
  - Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong
  - Zhongshan Hospital Fudan University, Guangdong Province, Shanghai Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- Centro Comprensivo de Cancer de UPR, San Juan, Puerto Rico
- National Cancer Centre Singapore, Singapore, Singapore
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Chang Gung Hospital-Lin Kou Medical Center, Taoyuan District